CLINICAL TRIAL: NCT02634567
Title: Attention/Working Memory Rehabilitation in Multiple Sclerosis: A Pilot Project Using Cogmed Working Memory Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Sarah Morrow, MD, MS, FRCPC (Neurology), London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 107343
Record Dates: First submitted 2015-12-11; First posted 2015-12-18 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Treatment as Usual (No Intervention): This group will not any training with the Cogmed training program.
- Training Group (Experimental): This group will receive intervention with the Cogmed training program and coach over a period of 5 weeks.
  Interventions: Behavioral: Cogmed Working Memory Training (CWMT)

INTERVENTIONS:
Behavioral: Cogmed Working Memory Training (CWMT) — The CWMT (Cogmed) method consists of 25 training sessions done online. Each participant assigned to the training group will complete eight exercises for five weeks with five sessions every week. Each session consists of a selection of various tasks that target the different aspects of attention/working memory. Participants will engage in weekly discussions over the phone for about 1 hour with an assigned Cogmed coach who will provide support and encouragement over the 5 weeks.
  Arms: Training Group

SUMMARY:
Patients diagnosed with any type of multiple sclerosis (MS) who show objective evidence of attention problems will be randomized to standard medical care (treatment as usual) or attention training, which will be completed at their home using a commercially available attention training task (Cogmed Working Memory Training - CWMT) for 5 weeks. Patients will undergo cognitive testing before and after intervention and at 6 months follow up.

DETAILED DESCRIPTION:
MS patients who meet the inclusion criteria of the study showing deficits on at least 2 of 3 attention/working measures who will then be randomized to either a treatment group (cognitive rehabilitation training) or a control group (standard clinical care). Patients must show mild to moderate-severe impairment on 2 out of 3 test measures of processing speed and sustained attention to be included in the study. Participants will undergo cognitive testing (Minimal Assessment of Cognitive Function in MS [MACFIMS] performed at Dr. Morrow's cognitive clinic at Parkwood Hospital) at pre- and post-treatment, and also at 6-months follow-up. Participants will also fill out non-cognitive measures in the form of questionnaires regarding quality of life (QoL), self-efficacy, stress, and copying strategies at both pre and post treatment. In addition, the intervention group will undergo attention training using CWMT for 5 days per week (30-45 minutes daily) for 5 weeks. They will complete this training by themselves in their home. The assigned Cogmed coach will set up the Cogmed program for the duration of the trail on the training group participant's computers. The study will not be able to continue to pay for the Cogmed program after the 5 week training sessions. Participants are welcome to purchase the software themselves after the entire study has ended if they would like at: http://www.cogmed.com/. The CWMT (Cogmed) method consists of 25 training sessions done online. Each participant assigned to the training group will complete eight exercises for five weeks with five sessions every week. The Cogmed program uses an adaptive training approach in which the difficulty level of the training is adjusted in real time (trial by trial basis) based on the trainee's performance. Each session consists of a selection of various tasks that target the different aspects of attention/working memory. Specifically, each session will involve training on visuospatial working memory tasks (e.g., remembering the position of objects in a 4 x 4 Grid) as well as verbal working memory tasks (e.g., remembering phonemes, letters, or digits). Given that adults will be involved in this study, Cogmed QM will be used, a version of the CWMT program adapted for adults. Participants will engage in weekly discussions over the phone for about 1 hour with an assigned Cogmed coach who will provide support and encouragement over the 5 weeks. Additional calls will be made if the Cogmed coaches see the participant is not completing their online training. Each participant will be assigned a Cogmed qualified coach who is responsible for providing structure, motivation, and feedback on training progress in order to optimize training gains. Before Cogmed training begins, each participant in the training group will be visited once by their respective Cogmed coach who will ensure that participants' daily Cogmed sessions will be conducted in a space in their home that is conducive to attention training (e.g., little clutter, private area of the home) and ensure consistency between participants. During training, each participant's performance will be tracked online and will be reviewed by the participant and his/her coach in weekly telephone meetings throughout the five week period. The participant's performance will be tracked online on the Cogmed platform. The Cogmed coaches set up the program for the participants and assign them a username. The Cogmed coaches can track the individual's performance and see who has completed the training based on their username. No Internet Protocol (IP) information will be collected. At the end of training, the coach will summarize the training by telephone with the participant.

ELIGIBILITY:
Gender Both: both female and male participants are being studied

Age Limits Minimum Age: 18 years Maximum Age: 64 years

Accepts Healthy Volunteers? No

Eligibility Criteria

Inclusion Criteria:

* Males/Females, Ages 18-64, with any type of MS
* Lower to moderate physical disability
* Demonstrated impaired attention/working memory on 2 of 3 measures (Patients with a z-score lower than -1.5 on at least 2 of the 3 measures will be characterized as showing attention/working memory deficits)
* Patients must have a Mac or personal computer (PC) computer at home with access to the internet

Exclusion Criteria:

* Clinical relapse/steroid treatment 1 month prior to study entry
* Physical disability that prevents completion of study measures or training
* History of severe mental illness or daily marijuana use
* Those who do not meet the inclusion criteria.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-04; Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Paced Auditory Serial Addition Test | 7 months
  Cognitive test; Change pre- to post-test between groups
Symbol Digit Modalities Test | 7 months
  Cognitive test; Change pre- to post-test between groups
Stroop colour word test | 7 months
  Cognitive test; Change pre- to post-test between groups

SECONDARY OUTCOMES:
Judgement of Line Orientation | 7 months
  Cognitive test; Change pre- to post-test between groups
Controlled Oral Word Association Test | 7 months
  Cognitive test; Change pre- to post-test between groups
California Verbal Learning Test | 7 months
  Cognitive test; Change pre- to post-test between groups
Brief Visual Memory Test | 7 months
  Cognitive test; Change pre- to post-test between groups
Delis-Kaplan Executive Function System Sorting Test | 7 months
  Cognitive test; Change pre- to post-test between groups
Beck Depression Inventory - Fast Screen | 7 months
  Non-cognitive Questionnaire; Change pre- to post-test between groups
Hospital Anxiety and Depression Scale | 7 months
  Non-cognitive Questionnaire; Change pre- to post-test between groups
Fatigue Severity Scale | 7 months
  Non-cognitive Questionnaire; Change pre- to post-test between groups
Short Form Health Survey | 7 months
  Non-cognitive Questionnaire; Change pre- to post-test between groups
Dysexecutive Questionnaire | 7 months
  Non-cognitive Questionnaire; Change pre- to post-test between groups in terms of the amount of self-reported issues with executive functions.
Cognitive Failures Questionnaire | 7 months
  Non-cognitive Questionnaire; Change pre- to post-test between groups in terms of the amount of self-reported cognitive issues
BRIEF Cope | 7 months
  Non-cognitive Questionnaire; Change pre- to post-test between groups
Social Stress and Support Interview | 7 months
  Non-cognitive Questionnaire; Change pre- to post-test between groups
Multiple Sclerosis Neuropsychological Screening Questionnaire | 7 months
  Non-cognitive Questionnaire; Change pre- to post-test between groups
Perceived Deficits Questionnaire | 7 months
  Non-cognitive Questionnaire; Change pre- to post-test between groups
Visual Spatial Span Board Assessment | 7 months
  Cognitive Test; Change pre- to post-test between groups in the amount of correct sequencing of repeated taping blocks in forward or reverse order from sequence presented by the examiner.
Digit Span | 7 months
  Cognitive Test; Change pre- to post-test between groups in terms of digit sequence memorized and repeated. A span of 3-9 digits will be repeated forwards and backwards after presentation from the examiner.
Arithmetic | 7 months
  Cognitive Test; Change pre- to post-test between groups, elementary math presented and solved without a pencil and paper.
Letter-Number Sequencing | 7 months
  Cognitive Test; Change pre- to post-test between groups, presented with a combination of letters and numbers; must repeat numbers in ascending order and letters in alphabetical order to examiner.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Morrow, MD, MS, FRCPC (Neurology), Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada